CLINICAL TRIAL: NCT02322840
Title: An Initial Evaluation of the Safety and Performance of the Transcatheter Mitral Intrepid Valve Replacement System in Patients With Severe, Symptomatic Mitral Regurgitation
Brief Title: Transcatheter Mitral Valve Replacement System (TMVR) Pilot Study and The Early Feasibility Study of the TMVR Transseptal System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-1403 & MDT19042TMV002
Record Dates: First submitted 2014-10-31; First posted 2014-12-23 (Estimated); Results first posted 2025-11-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcatheter Mitral Valve Replacement (TMVR) Implant (Experimental): Twelve TMVR Implant
  Interventions: Device: Twelve TMVR Implant; Device: Medtronic Intrepid™ Transcatheter Transfemoral Mitral Valve Replacement System

INTERVENTIONS:
Device: Twelve TMVR Implant — Implantation of the Twelve TMVR System - Apical
  Other Names: Medtronic Intrepid™ Transcatheter Mitral Valve Replacement System
Device: Medtronic Intrepid™ Transcatheter Transfemoral Mitral Valve Replacement System — Implantation of the Medtronic Intrepid™ Transcatheter Mitral Valve- Transfemoral
  Other Names: Medtronic Intrepid™ Transcatheter Mitral Valve Replacement System

SUMMARY:
PILOT:

The study is a pilot trial to evaluate the safety and performance of the Twelve TMVR System in high risk mitral regurgitation patients.

EFS:

The study is an Early Feasibility Study to evaluate the safety and performance of the Medtronic Intrepid™ Transcatheter Mitral Valve Replacement System with Transfemoral Transseptal access in Patients with moderate-Severe or severe, Symptomatic Mitral Regurgitation

DETAILED DESCRIPTION:
PILOT:

The study is a prospective, multi-center, non-randomized study to evaluate the safety and performance of The Intrepid™ TMVR System in patients with severe, symptomatic mitral regurgitation, who are at high risk for conventional mitral valve surgery.

EFS:

The study is a multi-center, prospective, non-randomized, trial to evaluate the safety and performance of the Medtronic Intrepid™ Transcatheter Mitral Valve Replacement System with Transfemoral Transseptal access in Patients with Moderate-Severe or Severe, Symptomatic Mitral Regurgitation

ELIGIBILITY:
Key Inclusion Criteria:

* Severe mitral regurgitation (PILOT)
* moderate-severe or severe mitral regurgitation (EFS)
* Symptomatic mitral regurgitation (NYHA Class II-IV)
* Deemed to be at high risk for conventional mitral valve surgery by the local heart team (including, at minimum, a cardiac surgeon, interventional cardiologist, and an echocardiologist) (PILOT and EFS)
* Subjects anatomically suitable for the Intrepid TMVR delivery system, including transfemoral and transseptal access (EFS only)
* Native mitral valve geometry and size compatible with the Intrepid™ TMVR (PILOT)

Key Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 20 (PILOT) or <30% (EFS)
* Evidence of intracardiac mass, thrombus, or vegetation
* Prior valve surgery or need for other valve surgery
* Prior stroke within 30 days (PILOT) or 90 days (EFS)
* Gastrointestinal bleeding within 6 months (PILOT)
* Prior myocardial infarction 90 days (EFS)
* Need for coronary revascularization
* History of, or active, endocarditis if antibiotics are required (EFS)
* Renal insufficiency; Serum Creatinine > 2.5 mg/dL (PILOT) or Creatinine Clearance <30 cc/min (EFS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnett Stahl, Study Director — Medtronic
Locations (32):
- United States (21):
  - Abrazo Arizona Heart Hospital - EFS, Phoenix, Arizona
  - Cedars-Sinai Medical Center - PILOT, Los Angeles, California
  - Piedmont Atlanta Hospital - PILOT, Atlanta, Georgia
  - Northwestern Memorial Hospital - PILOT, Chicago, Illinois
  - University of Michigan Health System - University Hospital - PILOT, Ann Arbor, Michigan
  - Corewell Health - EFS, Grand Rapids, Michigan
  - Abbott Northwestern Hospital - EFS, Minneapolis, Minnesota
  - Abbott Northwestern Hospital - PILOT, Minneapolis, Minnesota
  - Barnes Jewish Hospital - PILOT, St Louis, Missouri
  - NYU Langone Medical Center - PILOT, New York, New York
  - The Mount Sinai Hospital (New York NY) - EFS, New York, New York
  - The Mount Sinai Hospital (New York NY) - PILOT, New York, New York
  - New York-Presbyterian Hospital Columbia University Medical Center - EFS, New York, New York
  - New York-Presbyterian Hospital Columbia University Medical Center - PILOT, New York, New York
  - Oregon Health & Science University Hospital - EFS, Portland, Oregon
  - UPMC Pinnacle Harrisburg Campus - EFS, Wormleysburg, Pennsylvania
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital - PILOT, Dallas, Texas
  - Houston Methodist Hospital - PILOT, Houston, Texas
  - University of Virginia Medical Center - EFS, Charlottesville, Virginia
  - Aurora Saint Luke's Medical Center - EFS, Milwaukee, Wisconsin
  - Aurora Saint Lukes Medical Center - PILOT, Milwaukee, Wisconsin
- Australia (3):
  - Monash Health - PILOT, Clayton, Victoria
  - The Alfred Hospital - PILOT, Melbourne
  - Royal Prince Alfred Hospital - PILOT, Sydney
- Rigshospitalet - PILOT, Copenhagen, Denmark
- Helsinki University Hospital - PILOT, Helsinki, Finland
- France (2):
  - Centre Hospitalier Régional Universitaire de Lille - PILOT, Lille
  - Clinique Pasteur - PILOT, Toulouse
- Hygeia Hospital - PILOT, Athens, Greece
- United Kingdom (3):
  - Royal Sussex County Hospital - PILOT, Brighton
  - The Leeds Teaching Hospitals NHS Trust - Leeds General Infirmary - PILOT, Leeds
  - Guys & St Thomas NHS Foundation Trust - St Thomas Hospital - PILOT, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang GHL, Rajagopal V, Sorajja P, Bajwa T, Gooley R, Walton A, Modine T, Ng MK, Williams MR, Zajarias A, Hildick-Smith D, Tchetche D, Spargias K, Rajani R, Bapat VN, De Backer O, Blackman D, McCarthy P, Laine M, Jain R, Martin R, Thaden JJ, Marka NA, Mack M, Adams DH, Leon MB, Reardon MJ. Five-year outcomes of the early-generation Intrepid transapical transcatheter mitral valve replacement system. EuroIntervention. 2026 Feb 2;22(3):e172-e182. doi: 10.4244/EIJ-D-25-01133. PMID 41251714
- [Derived] Zahr F, Song HK, Chadderdon SM, Gada H, Mumtaz M, Byrne T, Kirshner M, Bajwa T, Weiss E, Kodali S, George I, Heiser J, Merhi WM, Thaden JJ, Zhang A, Lim DS, Reardon MJ, Adams DH, Mack MJ, Leon MB. 30-Day Outcomes Following Transfemoral Transseptal Transcatheter Mitral Valve Replacement: Intrepid TMVR Early Feasibility Study Results. JACC Cardiovasc Interv. 2022 Jan 10;15(1):80-89. doi: 10.1016/j.jcin.2021.10.018. Epub 2021 Nov 6. PMID 34747699
- [Derived] Bapat V, Rajagopal V, Meduri C, Farivar RS, Walton A, Duffy SJ, Gooley R, Almeida A, Reardon MJ, Kleiman NS, Spargias K, Pattakos S, Ng MK, Wilson M, Adams DH, Leon M, Mack MJ, Chenoweth S, Sorajja P; Intrepid Global Pilot Study Investigators. Early Experience With New Transcatheter Mitral Valve Replacement. J Am Coll Cardiol. 2018 Jan 2;71(1):12-21. doi: 10.1016/j.jacc.2017.10.061. Epub 2017 Nov 16. PMID 29102689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred April 2015 to March 2019 at 23 sites (12 U.S.,3 Australia, 8 Europe)(PILOT), Jan. 2020 to Aug. 2022 at 11 U.S sites (EFS). Patients with severe, symptomatic mitral regurgitation at high surgical risk (PILOT) or moderate-severe or severe, symptomatic mitral regurgitation, ineligible for conventional mitral valve surgery (EFS) were screened for eligibility, provided informed consent, met all inclusion criteria, and no exclusion criteria, were enrolled.
Pre-assignment Details: These are single-arm studies. Patients who signed informed consent & fulfill inclusion criteria and none of the exclusion criteria listed below are eligible for enrollment. A Patient Review Committee (PRC) (PILOT)/ Screening Committee (EFS), which consisted of cardiac surgery, interventional cardiology, and echocardiology representatives who were not participating investigators, reviewed potential patients' clinical and imaging data to help ensure appropriate patient selection across all sites.
Groups:
- Transcatheter Mitral Valve Replacement (TMVR) Implant: Twelve TMVR Implant
  Twelve TMVR Implant: Implantation of the Twelve TMVR System -Apical
  Medtronic Intrepid™ Transcatheter Transfemoral Mitral Valve Replacement System: Implant of Intrepid valve -Transfemoral
Period: Overall Study
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Started | 128 (95 (PILOT) 33 (EFS))
Completed | 58 (27 (PILOT) 31 (EFS))
Not Completed | 70

BASELINE CHARACTERISTICS:
Population: 95 (PILOT) 33 (EFS)
Groups:
- Transcatheter Mitral Valve Replacement (TMVR) Implant: Twelve TMVR Implant: Implantation of the Twelve TMVR System -Apical
  Medtronic Intrepid™ Transcatheter Transfemoral Mitral Valve Replacement System: Implant of Intrepid valve -Transfemoral
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] — PILOT Population: PILOT
  years
    number analyzed (Participants) | 95
    (all) | 74.0 (9.2)
Age, Continuous [Mean (Standard Deviation); unit: years] — EFS Population: EFS
  years
    number analyzed (Participants) | 33
    (all) | 78.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: PILOT
  Participants
    number analyzed (Participants) | 95
    Female | 41
    Male | 54
Sex: Female, Male [Count of Participants; unit: Participants] — Population: EFS
  Participants
    number analyzed (Participants) | 33
    Female | 12
    Male | 21
Race/Ethnicity, Customized [Number; unit: Paticipants] — PILOT Population: PILOT
  Paticipants
    Caucasian: number analyzed (Participants) | 95
    Caucasian | 81
    Hispanic or Latino: number analyzed (Participants) | 95
    Hispanic or Latino | 3
    Black or African American: number analyzed (Participants) | 95
    Black or African American | 9
    Asian: number analyzed (Participants) | 95
    Asian | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — EFS Population: Data not collected for EFS participants
Region of Enrollment [Count of Participants; unit: Participants] — Population: PILOT
  Participants
    Greece: number analyzed (Participants) | 95
    Greece | 3
    United States: number analyzed (Participants) | 95
    United States | 52
    Denmark: number analyzed (Participants) | 95
    Denmark | 2
    United Kingdom: number analyzed (Participants) | 95
    United Kingdom | 9
    Australia: number analyzed (Participants) | 95
    Australia | 19
    France: number analyzed (Participants) | 95
    France | 9
    Finland: number analyzed (Participants) | 95
    Finland | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: EFS
  Participants
    United States: number analyzed (Participants) | 33
    United States | 33
STS Score - PROM (MV Replacement Only) [Mean (Standard Deviation); unit: % risk of mortality] — STS-PROM= Society of Thoracic Surgeons Predictive Risk of Mortality
  STS-PROM score is a tool developed by the Society of Thoracic Surgeons to estimate a patients risk of death after cardiac surgery. The model incorporates a range of factors such as patient demographics, comorbidities, physiological data and procedure information that influence a patient risk. Population: PILOT
  % risk of mortality
    number analyzed (Participants) | 95
    (all) | 6.5 (4.8)
STS Score- PROM (MV Replacement only) [Mean (Standard Deviation); unit: % risk of mortality] — STS-PROM= Society of Thoracic Surgeons Predictive Risk of Mortality
  STS-PROM score is a tool developed by the Society of Thoracic Surgeons to estimate a patients risk of death after cardiac surgery. The model incorporates a range of factors such as patient demographics, comorbidities, physiological data and procedure information that influence a patient risk. Population: EFS
  % risk of mortality
    number analyzed (Participants) | 33
    (all) | 5.3 (2.8)
Creatinine Clearance [Mean (Standard Deviation); unit: cc/min] — Population: PILOT One subject had a serum creatinine level deemed below the plausible lower threshold by our medical expert (<0.4 mg/dL) and was therefore excluded from the analysis.
  cc/min
    number analyzed (Participants) | 94
    (all) | 60.3 (25.0)
Creatinine Clearance [Mean (Standard Deviation); unit: cc/min] — Population: EFS
  cc/min
    number analyzed (Participants) | 33
    (all) | 61.4 (25.7)
NYHA Class [Count of Participants; unit: Participants] — NYHA is measured by the patients physical activity limitations and places the patients in one of four classes.
  NYHA Class I is measured by no limitations of physical activity. NYHA Class II is measured by slight limitations of physical activity. NYHA Class III is measured by marked limitation of physical activity. NYHA Class IV is measured by symptoms of heart failure at rest. Any physical activity causes discomfort. Population: PILOT
  Participants
    number analyzed (Participants) | 95
    NYHA I | 0.0
    NYHA II | 11
    NYHA III | 71
    NYHA IV | 13
NYHA Class [Count of Participants; unit: Participants] — NYHA is measured by the patients physical activity limitations and places the patients in one of four classes.
  NYHA Class I is measured by no limitations of physical activity. NYHA Class II is measured by slight limitations of physical activity. NYHA Class III is measured by marked limitation of physical activity. NYHA Class IV is measured by symptoms of heart failure at rest. Any physical activity causes discomfort. Population: EFS
  Participants
    number analyzed (Participants) | 33
    NYHA l | 0
    NYHA ll | 10
    NYHA lll | 22
    NYHA lV | 1
Previous Myocardial infarction [Count of Participants; unit: Participants] — Population: PILOT
  Participants
    number analyzed (Participants) | 95
    (all) | 40
Previous Myocardial infarction [Count of Participants; unit: Participants] — Population: EFS
  Participants
    number analyzed (Participants) | 33
    (all) | 9
Previous Cardiovascular Surgery [Count of Participants; unit: Participants] — Population: PILOT
  Participants
    number analyzed (Participants) | 95
    (all) | 45
Previous Cardiovascular Surgery [Count of Participants; unit: Participants] — Population: EFS
  Participants
    number analyzed (Participants) | 33
    (all) | 16
Mitral Valve Etiology [Count of Participants; unit: Participants] — Mitral Regurgitation is blood flowing backward through the mitral valve.
  Primary Mitral Regurgitation is measured by a problem with the mitral valve apparatus itself.
  Secondary Mitral regurgitation is measured by an enlarged or weakened left side of the heart that pulls the valve leaflets apart and prevents them from closing. The mitral valve structure is normal. Population: PILOT One subject did not have either Core lab nor Site reported MR Etiology
  Participants
    number analyzed (Participants) | 94
    Primary | 20
    Secondary | 74
Mitral Valve Etiology [Count of Participants; unit: Participants] — Mitral Regurgitation is blood flowing backward through the mitral valve.
  Primary Mitral Regurgitation is measured by a problem with the mitral valve apparatus itself.
  Secondary Mitral regurgitation is measured by an enlarged or weakened left side of the heart that pulls the valve leaflets apart and prevents them from closing. The mitral valve structure is normal. Population: EFS
  Participants
    number analyzed (Participants) | 33
    Primary | 20
    Secondary | 13
Atrial Fibrillation [Count of Participants; unit: Participants] — Population: PILOT
  Participants
    number analyzed (Participants) | 95
    (all) | 57
Atrial Fibrillation [Count of Participants; unit: Participants] — Population: EFS
  Participants
    number analyzed (Participants) | 32
    (all) | 15
EUROSCORE II (%) [Mean (Standard Deviation); unit: % risk of mortality] — Population: PILOT
  % risk of mortality
    number analyzed (Participants) | 95
    (all) | 8.0 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Adverse Events
Description: PILOT: Site Reported Serious Adverse Events Implant or Delivery Related Through 30-Days EFS: Implant, Delivery or device related serious adverse events through 30 days post procedure
Time Frame: 30 days
Population: PILOT: 95 participants EFS: 33 participants
Measure: Number; unit: % of subjects with Event
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 128
% of subjects with Event
  PILOT: number analyzed (Participants) | 95
  PILOT | 67
  EFS Implant or Delivery Related: number analyzed (Participants) | 33
  EFS Implant or Delivery Related | 72.7
  EFS Device Related: number analyzed (Participants) | 33
  EFS Device Related | 36.4

2. Secondary Outcome: Number of Subjects With Procedural Success
Description: PILOT: Successful access, delivery of implant, and retrieval of the delivery system EFS: Successful access, delivery of implant, and retrieval of the delivery system
Time Frame: Procedure
Population: PILOT: One subject had their procedure aborted prior to delivery catheter insertion and was thus excluded from deployment and retrieval denominator
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 128
Participants
  PILOT: Successful access: number analyzed (Participants) | 95
  PILOT: Successful access | 94
  PILOT: Successful Delivery of implant: number analyzed (Participants) | 94
  PILOT: Successful Delivery of implant | 90
  PILOT: Successful retrieval of the delivery system: number analyzed (Participants) | 94
  PILOT: Successful retrieval of the delivery system | 94
  EFS: Procedural Success (Number of Patients with Successful TMVR Placement): number analyzed (Participants) | 33
  EFS: Procedural Success (Number of Patients with Successful TMVR Placement) | 31

3. Secondary Outcome: Change in Mitral Regurgitation (MR) From Baseline Through 30 Days
Description: PILOT: Change in MR Grade from baseline measured by echo through 30 days post-procedure. Measured by Echo 30 days post procedure.
Time Frame: 30 days
Population: Number of subjects with evaluable baseline and 30 day CoreLab echo MR grading.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 71
Participants
  PILOT: Improved | 71
  PILOT: No change | 0
  PILOT: Worsened | 0

4. Secondary Outcome: Change in Mitral Regurgitation (MR) From Baseline Through 30 Days
Description: EFS: Change in MR Grade from Baseline measured by echo through 30 days post-procedure. Measured by Echo 30 days post procedure.
Time Frame: Through 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 30
Participants
  Improved | 30
  No change | 0
  Worsened | 0

5. Secondary Outcome: Change in New York Heart Association (NYHA) From Baseline Through 30 Days
Description: PILOT: Change in NYHA Class from Baseline through 30 days post-procedure.
Time Frame: Through 30 days
Population: PILOT: Number of subjects with evaluable baseline and 30 days NYHA classification.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 93
Participants
  Improved | 54
  No change | 20
  Worsened | 1
  Died Prior to Visit | 18

6. Secondary Outcome: Change in New York Heart Association (NYHA) From Baseline Through 30 Days
Description: EFS: Change in NYHA Class from Baseline through 30 days post procedure
Time Frame: Through 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 30
Participants
  Improved | 21
  No Change | 6
  Worsened | 3
  Died Prior to Visit | 0

7. Secondary Outcome: Number of Subjects Without Mitral Valve Stenosis
Description: PILOT: No significant mitral Valve (MV) Stenosis measured by echo through 30 days post-procedure EFS: No Significant Mitral Valve (MV) Stenosis measured by echo through 30 days post-procedure
Time Frame: Through 30 days
Population: PILOT: N= 62. Number of subjects with evaluable baseline and 30 day CoreLab echoes for MV stenosis; defined as an MV mean gradient < 5 mmHg and effective orifice area (EOA) ≥ 1.5 cm² based on echocardiography core lab data.
  EFS: N=25. Number of subjects with EOA >= 1.5 cm2, Transmitral Gradient <5 mmHg, PVL <=Mild, and No Hemolysis with PVL
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 87
Participants
  PILOT: number analyzed (Participants) | 62
  PILOT | 19
  EFS: number analyzed (Participants) | 25
  EFS | 11

8. Secondary Outcome: Number of Subject With Left Ventricle Output Tract (LVOT) Patency
Description: PILOT: LVOT patency measured by echo through 30 days post-procedure.
Time Frame: Through 30 days
Population: Number of subjects with evaluable baseline and 30 day CoreLab echoes for LVOT patency.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 65
Participants | 62

9. Secondary Outcome: Percent of Subject With Left Ventricular Outflow Tract (LVOT) Patency
Description: EFS: Left Ventricular Outflow Tract (LVOT) Patency measured by echo through 30 days post-procedure
Time Frame: 30 Days post procedure
Population: Number of subjects with evaluable baseline and 30 day CoreLab echoes for LVOT patency.
Measure: Number; unit: Percent
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 29
Percent | 100

10. Secondary Outcome: Number of Subjects With Greater Than or Equal Moderate (2+) Mitral Regurgitation at 30-days
Description: PILOT: Number of subjects with a core lab-evaluated mitral regurgitation grade greater than or equal to moderate at 30-days
Time Frame: Through 30 days
Population: Number of subjects with a core lab-evaluated mitral regurgitation grade greater than or equal to moderate at 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Transcatheter Mitral Valve Replacement (TMVR) Implant
Number analyzed (Participants) | 71
Participants | 0

ADVERSE EVENTS:
Time Frame: PILOT: Adverse event data was collected through 5 years for each participant EFS: Adverse event data was collected through 4 years.
Description: PILOT: MedDRA 25 EFS: MedDRA 26 All adverse events were adjudicated by CEC for seriousness and relatedness
Groups:
- PILOT: Twelve TMVR Implant: Implantation of the Twelve TMVR System -Apical (N=95)
- Early Feasibility Study (EFS): Medtronic Intrepid™ Transcatheter Transfemoral Mitral Valve Replacement System: Implant of Intrepid valve -Transfemoral (N=33)
Arm/Group | PILOT | Early Feasibility Study (EFS)
All-Cause Mortality (participants affected / at risk) | 62/95 | 7/33
Serious Adverse Events (participants affected / at risk) | 93/95 | 32/33
Other Adverse Events (participants affected / at risk) | 88/95 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PILOT (N=95) | Early Feasibility Study (EFS) (N=33)
Anaemia (Blood and lymphatic system disorders) | 14 (21) | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 5 (5) | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0
Acute left ventricular failure (Cardiac disorders) | 1 (2) | 0
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 0
Angina unstable (Cardiac disorders) | 1 (1) | 0
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0
Arrhythmia (Cardiac disorders) | 1 (1) | 0
Arrhythmic storm (Cardiac disorders) | 1 (1) | 0
Atrial fibrillation (Cardiac disorders) | 12 (13) | 0
Atrial flutter (Cardiac disorders) | 2 (2) | 0
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0
Atrial thrombosis (Cardiac disorders) | 2 (2) | 0
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0
Bundle branch block left (Cardiac disorders) | 1 (1) | 0
Cardiac arrest (Cardiac disorders) | 11 (11) | 0
Cardiac failure (Cardiac disorders) | 16 (28) | 0
Cardiac failure acute (Cardiac disorders) | 9 (12) | 0
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0
Cardiac failure congestive (Cardiac disorders) | 24 (37) | 0
Cardiac perforation (Cardiac disorders) | 1 (1) | 0
Cardiac pseudoaneurysm (Cardiac disorders) | 1 (1) | 0
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0
Cardiogenic shock (Cardiac disorders) | 12 (12) | 0
Cardiomyopathy (Cardiac disorders) | 3 (3) | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 0
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 0
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0
Left ventricular failure (Cardiac disorders) | 1 (1) | 0
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0
Myocardial infarction (Cardiac disorders) | 2 (2) | 0
Palpitations (Cardiac disorders) | 2 (2) | 0
Pericardial haemorrhage (Cardiac disorders) | 4 (4) | 0
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0
Tachycardia (Cardiac disorders) | 1 (1) | 0
Tricuspid valve incompetence (Cardiac disorders) | 2 (2) | 0
Ventricle rupture (Cardiac disorders) | 1 (1) | 0
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0
Ventricular fibrillation (Cardiac disorders) | 6 (7) | 0
Ventricular tachycardia (Cardiac disorders) | 12 (16) | 0
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1) | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0
Gastritis (Gastrointestinal disorders) | 1 (1) | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 0
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0
Asthenia (General disorders) | 2 (2) | 0
Cardiac death (General disorders) | 1 (1) | 0
Chest pain (General disorders) | 3 (3) | 0
Death (General disorders) | 1 (1) | 0
Multi-organ disorder (General disorders) | 1 (1) | 0
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 0
Pain (General disorders) | 1 (1) | 0
Physical deconditioning (General disorders) | 2 (2) | 0
Prosthetic cardiac valve stenosis (General disorders) | 1 (1) | 0
Prosthetic cardiac valve thrombosis (General disorders) | 1 (1) | 0
Pyrexia (General disorders) | 2 (2) | 0
Sudden cardiac death (General disorders) | 1 (1) | 0
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0
Appendicitis (Infections and infestations) | 1 (1) | 0
Arthritis infective (Infections and infestations) | 1 (2) | 0
Bacteraemia (Infections and infestations) | 2 (2) | 0
Bacteriuria (Infections and infestations) | 1 (1) | 0
Biliary sepsis (Infections and infestations) | 1 (1) | 0
Bronchitis (Infections and infestations) | 1 (1) | 0
Bursitis infective (Infections and infestations) | 1 (1) | 0
COVID-19 (Infections and infestations) | 3 (3) | 0
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0
Cellulitis (Infections and infestations) | 4 (6) | 0
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0
Cystitis (Infections and infestations) | 1 (1) | 0
Endocarditis (Infections and infestations) | 1 (1) | 0
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 0
Epididymitis (Infections and infestations) | 1 (1) | 0
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0
Herpes zoster (Infections and infestations) | 1 (1) | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 0
Influenza (Infections and infestations) | 1 (2) | 0
Lower respiratory tract infection (Infections and infestations) | 2 (4) | 0
Myocardiac abscess (Infections and infestations) | 1 (1) | 0
Perineal abscess (Infections and infestations) | 1 (1) | 0
Pneumonia (Infections and infestations) | 14 (19) | 0
Pneumonia aspiration (Infections and infestations) | 3 (3) | 0
Pneumonia serratia (Infections and infestations) | 1 (1) | 0
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0
Pyelonephritis (Infections and infestations) | 1 (1) | 0
Respiratory tract infection (Infections and infestations) | 1 (1) | 0
Sepsis (Infections and infestations) | 3 (4) | 0
Septic shock (Infections and infestations) | 4 (4) | 0
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 0
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0
Urinary tract infection (Infections and infestations) | 8 (11) | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0
Urosepsis (Infections and infestations) | 3 (3) | 0
Wound infection (Infections and infestations) | 1 (1) | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 5 (5) | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 (1) | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 6 (6) | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 (2) | 0
Blood creatinine increased (Investigations) | 1 (1) | 0
Cardiac output decreased (Investigations) | 2 (2) | 0
Ejection fraction decreased (Investigations) | 1 (1) | 0
Electrocardiogram QRS complex prolonged (Investigations) | 1 (1) | 0
Haemoglobin decreased (Investigations) | 3 (3) | 0
Heart rate increased (Investigations) | 1 (1) | 0
Staphylococcus test positive (Investigations) | 1 (1) | 0
White blood cell count increased (Investigations) | 1 (1) | 0
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0
Gout (Metabolism and nutrition disorders) | 3 (3) | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 (5) | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 0
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0
Embolic stroke (Nervous system disorders) | 1 (1) | 0
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0
Ischaemic stroke (Nervous system disorders) | 1 (2) | 0
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0
Syncope (Nervous system disorders) | 3 (3) | 0
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 0
Device breakage (Product Issues) | 1 (1) | 0
Device dislocation (Product Issues) | 5 (5) | 0
Prosthetic cardiac valve malfunction (Product Issues) | 1 (1) | 0
Confusional state (Psychiatric disorders) | 1 (1) | 0
Delirium (Psychiatric disorders) | 3 (3) | 0
Mental status changes (Psychiatric disorders) | 2 (2) | 0
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 (2) | 0
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0
Renal failure (Renal and urinary disorders) | 7 (7) | 0
Renal impairment (Renal and urinary disorders) | 2 (2) | 0
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0
Urethral caruncle (Renal and urinary disorders) | 1 (4) | 0
Urinary retention (Renal and urinary disorders) | 1 (1) | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0
Drug therapy (Surgical and medical procedures) | 1 (1) | 0
Endotracheal intubation (Surgical and medical procedures) | 1 (1) | 0
Exploratory operation (Surgical and medical procedures) | 1 (1) | 0
Mechanical ventilation (Surgical and medical procedures) | 1 (1) | 0
Renal replacement therapy (Surgical and medical procedures) | 1 (1) | 0
Toe amputation (Surgical and medical procedures) | 1 (1) | 0
Aortic stenosis (Vascular disorders) | 1 (1) | 0
Arterial disorder (Vascular disorders) | 1 (1) | 0
Arterial perforation (Vascular disorders) | 1 (1) | 0
Haematoma (Vascular disorders) | 1 (1) | 0
Haemodynamic instability (Vascular disorders) | 3 (3) | 0
Haemorrhage (Vascular disorders) | 3 (3) | 0
Hypotension (Vascular disorders) | 6 (6) | 0
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 0
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 0
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 (1)
Acquired left ventricle outflow tract obstruction (Cardiac disorders) | 0 | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 | 2 (2)
Angina pectoris (Cardiac disorders) | 0 | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 | 7 (18)
Atrial flutter (Cardiac disorders) | 0 | 3 (3)
Atrial thrombosis (Cardiac disorders) | 0 | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 | 1 (1)
Bradycardia (Cardiac disorders) | 0 | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 | 1 (1)
Cardiac failure (Cardiac disorders) | 0 | 4 (4)
Cardiac failure acute (Cardiac disorders) | 0 | 7 (8)
Cardiac failure chronic (Cardiac disorders) | 0 | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 | 8 (10)
Cardiac pseudoaneurysm (Cardiac disorders) | 0 | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 | 1 (2)
Cardiomyopathy (Cardiac disorders) | 0 | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 (1)
Systolic dysfunction (Cardiac disorders) | 0 | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 | 2 (2)
Ventricular dyssynchrony (Cardiac disorders) | 0 | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 (1)
Cataract (Eye disorders) | 0 | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1)
Colitis (Gastrointestinal disorders) | 0 | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 4 (5)
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1 (1)
Chest pain (General disorders) | 0 | 1 (1)
Prosthetic cardiac valve stenosis (General disorders) | 0 | 1 (1)
Prosthetic cardiac valve thrombosis (General disorders) | 0 | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 | 1 (1)
Acute endocarditis (Infections and infestations) | 0 | 1 (1)
Bacteraemia (Infections and infestations) | 0 | 1 (1)
COVID-19 (Infections and infestations) | 0 | 2 (2)
Cellulitis (Infections and infestations) | 0 | 1 (2)
Endocarditis (Infections and infestations) | 0 | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 | 1 (1)
Fungal peritonitis (Infections and infestations) | 0 | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 | 1 (1)
Peritonitis (Infections and infestations) | 0 | 1 (2)
Pneumonia (Infections and infestations) | 0 | 2 (2)
Pneumonia aspiration (Infections and infestations) | 0 | 1 (1)
Prosthetic valve endocarditis (Infections and infestations) | 0 | 2 (2)
Pulmonary sepsis (Infections and infestations) | 0 | 1 (2)
Sepsis (Infections and infestations) | 0 | 3 (4)
Septic shock (Infections and infestations) | 0 | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 | 1 (1)
Urinary tract infection (Infections and infestations) | 0 | 2 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 8 (8)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 (1)
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 4 (4)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 3 (3)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1 (1)
Ejection fraction decreased (Investigations) | 0 | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 (1)
International normalised ratio increased (Investigations) | 0 | 1 (1)
Pulse absent (Investigations) | 0 | 1 (1)
Transvalvular pressure gradient increased (Investigations) | 0 | 1 (1)
Troponin increased (Investigations) | 0 | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 | 2 (3)
Dementia (Nervous system disorders) | 0 | 1 (1)
Dysarthria (Nervous system disorders) | 0 | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 (1)
Seizure (Nervous system disorders) | 0 | 1 (1)
Seizure like phenomena (Nervous system disorders) | 0 | 1 (1)
Syncope (Nervous system disorders) | 0 | 1 (1)
Device dislocation (Product Issues) | 0 | 1 (1)
Prosthetic cardiac valve malfunction (Product Issues) | 0 | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 | 8 (10)
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 | 3 (3)
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 (1)
Polyuria (Renal and urinary disorders) | 0 | 1 (1)
Renal failure (Renal and urinary disorders) | 0 | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Medical device implantation (Surgical and medical procedures) | 0 | 1 (1)
Air embolism (Vascular disorders) | 0 | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 | 2 (2)
Hypertension (Vascular disorders) | 0 | 1 (1)
Hypotension (Vascular disorders) | 0 | 4 (4)
Hypovolaemic shock (Vascular disorders) | 0 | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 (1)
Shock (Vascular disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PILOT (N=95) | Early Feasibility Study (EFS) (N=33)
Anaemia (Blood and lymphatic system disorders) | 19 (21) | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 8 (8) | 0
Leukocytosis (Blood and lymphatic system disorders) | 10 (10) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16) | 0
Atrial fibrillation (Cardiac disorders) | 25 (27) | 0
Cardiac failure (Cardiac disorders) | 7 (7) | 0
Cardiac failure congestive (Cardiac disorders) | 10 (12) | 0
Ventricular tachycardia (Cardiac disorders) | 12 (13) | 0
Constipation (Gastrointestinal disorders) | 5 (5) | 0
Pyrexia (General disorders) | 7 (7) | 0
Lower respiratory tract infection (Infections and infestations) | 5 (8) | 0
Pneumonia (Infections and infestations) | 9 (10) | 0
Urinary tract infection (Infections and infestations) | 23 (38) | 0
Fall (Injury, poisoning and procedural complications) | 14 (15) | 0
Skin laceration (Injury, poisoning and procedural complications) | 6 (6) | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (9) | 0
Hypervolaemia (Metabolism and nutrition disorders) | 10 (10) | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0
Dizziness (Nervous system disorders) | 6 (6) | 0
Delirium (Psychiatric disorders) | 7 (8) | 0
Acute kidney injury (Renal and urinary disorders) | 27 (32) | 0
Renal impairment (Renal and urinary disorders) | 10 (11) | 0
Urinary retention (Renal and urinary disorders) | 5 (5) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 5 (7) | 0
Hypertension (Vascular disorders) | 8 (8) | 0
Hypotension (Vascular disorders) | 11 (12) | 0
Orthostatic hypotension (Vascular disorders) | 5 (5) | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 16 (17)
Acquired left ventricle outflow tract obstruction (Cardiac disorders) | 0 | 3 (4)
Atrial fibrillation (Cardiac disorders) | 0 | 3 (3)
Atrial flutter (Cardiac disorders) | 0 | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 | 3 (3)
Bundle branch block left (Cardiac disorders) | 0 | 3 (3)
Cardiac failure (Cardiac disorders) | 0 | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 0 | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 | 4 (4)
Palpitations (Cardiac disorders) | 0 | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 0 | 4 (4)
Ventricular extrasystoles (Cardiac disorders) | 0 | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 0 | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 (2)
Asthenia (General disorders) | 0 | 2 (3)
Physical deconditioning (General disorders) | 0 | 2 (2)
Prosthetic cardiac valve thrombosis (General disorders) | 0 | 2 (2)
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 2 (2)
COVID-19 (Infections and infestations) | 0 | 9 (10)
Cystitis (Infections and infestations) | 0 | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 | 2 (2)
Urinary tract infection (Infections and infestations) | 0 | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 0 | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 | 4 (4)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 | 3 (3)
Vascular access site discharge (Injury, poisoning and procedural complications) | 0 | 2 (2)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 7 (8)
Anticoagulation drug level above therapeutic (Investigations) | 0 | 2 (2)
Anticoagulation drug level below therapeutic (Investigations) | 0 | 2 (2)
Ejection fraction decreased (Investigations) | 0 | 7 (7)
Free haemoglobin (Investigations) | 0 | 2 (2)
Transvalvular pressure gradient increased (Investigations) | 0 | 2 (2)
Troponin increased (Investigations) | 0 | 6 (7)
Weight increased (Investigations) | 0 | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 (4)
Dizziness (Nervous system disorders) | 0 | 3 (3)
Presyncope (Nervous system disorders) | 0 | 2 (2)
Prosthetic cardiac valve malfunction (Product Issues) | 0 | 2 (2)
Delirium (Psychiatric disorders) | 0 | 2 (2)
Depression (Psychiatric disorders) | 0 | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 | 11 (13)
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 (2)
Dysuria (Renal and urinary disorders) | 0 | 2 (2)
Haematuria (Renal and urinary disorders) | 0 | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Haematoma (Vascular disorders) | 0 | 2 (2)
Hypertension (Vascular disorders) | 0 | 4 (5)
Hypotension (Vascular disorders) | 0 | 4 (4)
Orthostatic hypotension (Vascular disorders) | 0 | 2 (2)
Peripheral venous disease (Vascular disorders) | 0 | 2 (2)

LIMITATIONS AND CAVEATS:
NCT02322840 covers the PILOT study and the Early Feasibility Study (EFS)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
According to the protocol, at the conclusion of the TMVR Pilot Study, a multi-center manuscript will be prepared for publication in a reputable scientific journal. The publication of the principal results from any single site experience within the study is not allowed until the preparation and publication of the multicenter results. Any follow-up publications would require prior written approval by the Publications Review Committee and the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT02322840/Prot_SAP_001.pdf